CLINICAL TRIAL: NCT04751565
Title: Analysis of the Treatment of Non-surgical Peri-implant Mucositis Treatment in Patients With Tissue-level (TL) and Bone-level (BL) Implants
Brief Title: Non Surgical Peri-implant Mucositis Treatment in Patients With Tissue-level and Bone-level Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Researcher, University of Messina
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-18/18
Record Dates: First submitted 2021-02-06; First posted 2021-02-12 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Intervention Model Description: Compare resolution of inflammation of naturally-occurring peri-implant mucositis (PM) at tissue-level (TL) and bone-level (BL) implants after non-surgical mechanical debridement.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue level implant Group (Experimental): Evaluation of healing of peri-implant mucositis after non-surgical supra and subgingival debridement in patients with tissue level implant
  Primary outcome
  The primary outcome will be based on probing depth (PD)
  Interventions: Other: Bleeding on Probing change reduction following peri-implant mucositis non surgical therapy
- Bone level implant Group (Experimental): Evaluation of healing of peri-implant mucositis after non-surgical supra and subgingival debridement in patients with bone level implant
  Primary outcome
  The primary outcome will be the change in Bleeding on Probing (BOP) (Lang, Joss, Orsanic, Gusberti, Siegrist, 1986).
  Interventions: Other: Bleeding on Probing change reduction following peri-implant mucositis non surgical therapy

INTERVENTIONS:
Other: Bleeding on Probing change reduction following peri-implant mucositis non surgical therapy — Statistically significant different in terms of Bleeding on Probing will be recorded between groups.

SUMMARY:
This study is designed to compare the resolution of inflammation of naturally-occurring peri-implant mucositis (PM) at tissue-level (TL) and bone-level (BL) implants after non-surgical mechanical debridement.

DETAILED DESCRIPTION:
Group A: Peri-implant mucositis (PM) at tissue-level (TL) implants after non-surgical mechanical debridement.

Group B: Peri-implant mucositis (PM) bone-level (BL) implants after non-surgical mechanical debridement.

ELIGIBILITY:
Inclusion criteria:

* Male and female aged > 18 years
* TL and BL titanium implants with smooth necks supporting cemented or screw-retained single-unit crowns diagnosed with PM (Berglundh, et al.,2018)
* Implants placed in both arches
* Patients with gingivitis or treated periodontitis (i.e., absence of residual PD > 5 mm)
* Presence of at least 2 mm of keratinized mucosa at implant sites.

Exclusion criteria:

* presence of medical conditions contraindicating treatment of peri-implant mucositis,
* regular use of anti-inflammatory drugs or antibiotics within 3 months prior to study enrollment

  * Presence of systemic diseases
  * Pregnant and lactating females
  * Smokers > 10 cigarettes/day
  * Use of inflammatory drugs or antibiotics within 3 months prior to study recruitment
  * Implants with modified (i.e. micro-rough) necks
  * Interproximal open contacts between implant restoration and adjacent teeth
  * Peri-implantitis (Renvert, et al., 2018)

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Bleeding on Probing (BOP) changes | Baseline (T0), 3-months (T1) and at 6-months (T2)
  Changes over time in BOP changes (percentage)

SECONDARY OUTCOMES:
Full mouth plaque score (FMPS) changes | Baseline (T0), 3-months (T1) and at 6-months (T2)
  Chenges in Full mouth plaque score (FMPS) (parameter)

OTHER OUTCOMES:
Pocket probing depth (PD) mm changes | Baseline (T0), 3-months (T1) and at 6-months (T2)
  changes in Pocket probing depth (PD)
Presence of plaque at implant sites according to plaque index (PlI) | Baseline (T0), 3-months (T1) and at 6-months (T2)
  Changes in presence of plaque at implant sites according to plaque index (PlI)

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Principal Investigator — Università degli Studi di Mesina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing study results
Supporting Information: Study Protocol
Time Frame: 6-months
Access Criteria: Pubmed website